CLINICAL TRIAL: NCT06562790
Title: A Phase 1, Randomised, Active-controlled, Blinded, Dose-ranging Study of the Safety, Tolerability, and Immunogenicity of an Inactivated Whole-cell Pneumococcal Vaccine (Gamma-PN3) in Elderly Participants
Brief Title: Study of Gamma PN3 in the Elderly
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GPN Vaccines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GPNV-006
Record Dates: First submitted 2024-08-18; First posted 2024-08-20 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2024-08

CONDITIONS: Pneumonia, Pneumococcal
MeSH Terms: conditions — Pneumonia, Pneumococcal | interventions — Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gamma-PN3 (Experimental): 2 doses on Days 1 and 29
  Interventions: Biological: Gamma PN3
- Prevnar (Active Comparator): 1 dose on Day 1 and saline placebo on Day 29.
  Interventions: Biological: Prevnar

INTERVENTIONS:
Biological: Gamma PN3 — 500, 1000 or 1500 µg by IM injection on Days 1 and 29
  Arms: Gamma-PN3
Biological: Prevnar — 1 dose on Day 1 and saline placebo on Day 29
  Arms: Prevnar

SUMMARY:
Phase 1 double- blind randomised active comparator dose escalating study of Gamma PN3 in the elderly

DETAILED DESCRIPTION:
The study is a phase 1, randomised, active-controlled, double-blind sequential ascending-dose study to evaluate the safety, tolerability, and immunogenicity of Gamma-PN3 in elderly adults. Three sequential, ascending dose cohorts are planned, with 35 participants per cohort randomised to one of two treatment arms. Administration of allocated study treatments will be on Days 1 and 29, with one treatment arm consisting of two doses of Gamma-PN3, and the treatment arm consisting of the comparator vaccine Prevenar 13® (one dose only, with second dose of Placebo).

Immunogenicity will be assessed at Day 29 and Day 57

ELIGIBILITY:
Inclusion Criteria:

1. Male or female volunteers aged 70 years and over at Screening.
2. In stable good general health as determined by the outcome of medical history, physical examination, and clinical judgement by the Investigator. Chronic stable non-inflammatory conditions such as hypertension, hyperlipidemia, well-controlled type 2 diabetes, stable asthma, controlled psychiatric conditions such as anxiety or depression, stable ischemic heart disease with heart failure not greater than NYHA Grade 1 and 2 are permitted, as determined by the Investigator.
3. Willing and able to give voluntary written informed consent before screening assessments commence.
4. Vital signs within the following ranges (inclusive):

   • Body temperature 35.5 to 37.7°C
   * Heart rate 50 to 100 beats per minute although atrial fibrillation is allowed.
   * Respiratory rate 12 to 22 breaths per minute
   * Systolic blood pressure 90 to 160 mmHg
   * Diastolic blood pressure 50 to 95 mmHg
5. 12-lead ECG parameters within the following ranges:

   • QTcB & QTcF - males ≤450 msec. females ≤470 msec
   * PR 100 to 240 msec inclusive
   * Heart rate (HR) 50 to 100 beats per minute (bpm) inclusive; atrial fibrillation is allowed.
6. Willing and able to communicate with the Investigator and study team and understands the requirements of the study.
7. Willing and able to undertake the study visits and all assessments, including possessing a suitable device and access to the internet for using the web-based electronic diary (e.g., smartphone, tablet, or computer) and able to use the device for this purpose.
8. Vaccinated against severe acute respiratory syndrome corona virus 2 (SARS-CoV-2; COVID-19) with a minimum of a prime and boost vaccinations.

Exclusion Criteria:

* 1. History of a previous Pneumovax 23® vaccination in last 12 months. 2. History of a previous Prevenar 13® or Prevenar 20® vaccination in last 12 months.

  3. Positive serology blood test for human immunodeficiency virus (HIV) antibodies, hepatitis B virus (HBV) surface antigen or Hepatitis C virus (HCV) antibodies. Positive serology to Hepatitis C due to previous successfully treated infection with negative polymerase chain reaction (PCR) is not exclusionary.

  4. Infectious disease including but not limited to COVID-19 and influenza within 30 days before Screening and any time between Screening and Day 1 first dose, as this may confound immune response to study vaccine.

  5. Liver function tests (including aspartate aminotransferase [AST], alanine aminotransferase [ALT], bilirubin) >1.5 upper limit of normal (ULN).

  6. Clinically significant abnormalities in laboratory tests (biochemistry, haematology), physical examination, or 12-lead ECG during the Screening period that, in the opinion of the Investigator, would affect immune response to vaccination and/or ability to fully participate in the study and/or not be in the individual's best interest to participate in the study. One re-test per abnormality is permitted.

  7. Participation in another clinical study of any investigational or licensed product (including investigational COVID-19 vaccines, drugs, medical devices) or medical procedure within 4 weeks from last study visit before screening.

  8. Plan to have a vaccine during the study period including COVID-19 booster. 9. Have had a live vaccine within three months of the first dose of study product or any other vaccine (including any COVID-19 vaccine) within 28 days of the first dose of study product.

Examples of live vaccines include, but are not limited to the following: measles, mumps, rubella, chicken pox/zoster (Zostavax; Shingrix is allowed), monkeypox, yellow fever, rabies, Bacillus Calmette-Guérin, and typhoid (oral) vaccines. Seasonal influenza vaccines for injection are generally killed virus vaccines and are permitted if administered at least 28 days before the first dose of study treatment and not during the enrollment or the study period. However, intranasal influenza vaccines are live attenuated vaccines and are not permitted within three months of first dose.

10. Have received blood or blood-derived products in the last three months before screening, which might interfere with assessment of the immune response.

11. Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the last six months before screening; or long-term systemic corticosteroid therapy (prednisone at a dose of 5mg daily or equivalent for more than two consecutive weeks within the last month before screening, depot or intraarticular steroids within 3 months before screening).

12. A systemic inflammatory condition such as rheumatoid arthritis or inflammatory bowel disease.

13. Any medical condition requiring immunosuppressive therapy. 14. History of severe allergic reaction e.g., severe cutaneous adverse reaction or anaphylaxis to any medicinal product or to any of the study treatments, including excipients.

15. Current alcohol abuse (> 21 U/week for men and 14 U/week for women), substance dependence including nicotine/tobacco smoking (defined as more than 5 cigarettes or tobacco/nicotine equivalent per day; smoking or vaping will not be permitted while at the study unit), any use of illicit drugs or other addiction which might interfere with the ability to comply with study procedures in the opinion of the Investigator; positive drugs of abuse screen (tricyclic antidepressants, opioids, and benzodiazepines are not exclusionary if prescribed by a physician and consistent with medical history) or positive alcohol breath test at Screening or pre-dose. One re-test permitted for drugs of abuse screen where justified (e.g., false positive suspected).

16. Clinically significant chronic illness that, in the opinion of the Investigator, is at a stage where it might interfere with study conduct or completion. Examples include congestive heart failure NHYA Grade 3 or 4, COAD with breathlessness interfering with daily activities; severe psychiatric conditions, poorly controlled asthma or diabetes 17. Any chronic medical condition e.g., asthma, gout, which is likely to need systemic corticosteroid therapy during the study.

18. Renal impairment requiring dialysis 19. Identified as a site employee of the Investigator or study center, with direct involvement in the proposed study or other studies under the direction of that Investigator or study center, as well as family members (i.e., immediate, husband, wife or de facto and their children, adopted or natural) of the site employees or the Investigator.

20. Poor venous access making scheduled blood sampling likely to be unsuccessful

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 105 (Actual)
Dates: Start 2024-08-26 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Adverse events | 57 days
  Spontaneous and diary recorded events
Geometric fold increase in IgG titre | 56 days
  Day 29 / Day 1 and Day 57/Day 1 geometric fold increase in IgG titre

SECONDARY OUTCOMES:
Geometric fold increase in OPA titre to 36 serotypes of S. pneumoniae | 56 days
  Day 29 / Day 1 and Day 57/Day 1 geometric fold increase in opsonophagocytic titre
Geometric fold increase in IgA | 56 days
  Day 29 / Day 1 and Day 57/Day 1 geometric fold increase in serum and mucosal IgA
Memory B cells | 56 days
  Memory B cell count
Rate of community acquired pneumonia | 1 year
  Number of participants with community acquired pneumonia

CONTACTS AND LOCATIONS:
Locations (1):
- CMAX Fusion, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No